CLINICAL TRIAL: NCT01419288
Title: Treadmill Training With Lower Extremity Amputees
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Eric Lamberg, Clinical Associate Professor, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0573-1
Record Dates: First submitted 2011-08-11; First posted 2011-08-18 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Traumatic Amputation of Lower Extremity
Keywords: Amputees

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Body weight support (Active Comparator)
  Interventions: Other: Treadmill Training
- Body weight support (Experimental)
  Interventions: Other: Treadmill Training

INTERVENTIONS:
Other: Treadmill Training — The program requires volunteer participants to attend 15 sessions over 10 to 12 weeks with a total time commitment of 13.5 hours. There is an initial testing session that includes an assessment of the participant's legs, balance, and walking abilities. The entire program includes 12 treadmill training visits that take place three times per week for four weeks, a post-training testing session one week after completion of the training, and a follow-up testing session four weeks after completion of the training.

SUMMARY:
Many people with a leg amputation have difficulty walking even after they have finished their rehabilitation. The purpose of this study is to see if a large amount of walking practice on a treadmill can improve functional abilities.

ELIGIBILITY:
Inclusion Criteria:

* Leg amputation that is either below the knee, through the knee, or above the knee
* Ability to walk with prosthetic
* Comfortably fitted with a prosthesis for at least 6 months
* Not currently receiving physical therapy for gait training
* Able to tolerate a moderate intensity exercise program

Exclusion Criteria:

* People with severe cardiac or pulmonary disease that limits ability to exercise.
* People with too much discomfort and/or pain that restricts their ability to walk.
* People with active wounds on their residual limb or contralateral foot.
* People who weigh more than 360lbs or are taller than 6'11" as the unweighing system can not support any greater load or height.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in 6-minute walk test | Baseline, after training, 1 month follow-up
  Participants will be assessed 3 times: Baseline, 1 week after completing the training protocol, and then 1 month after completing the training protocol

CONTACTS AND LOCATIONS:
Overall Officials: Eric Lamberg, EdD, PT, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University Medical Center, Stony Brook, New York, United States